CLINICAL TRIAL: NCT02929056
Title: A Prospective Randomized Comparative Parallel Study of Amniotic Membrane in the Management of Venous Leg Ulcerations
Brief Title: Amniotic Membrane Allograft Application in the Management of Venous Leg Ulcerations
Acronym: AmnioExCel
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: grant funding ended
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); BioDlogics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00059274
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Varicose Ulcer; Venous Insufficiency
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOC alginate dressing (Placebo Comparator): SOC absorptive alginate primary dressing in conjunction with a class II multi-layer compression wrap and standard debridement
  Interventions: Procedure: SOC alginate dressing and compression therapy
- AmnioExCel dressing (Experimental): AmnioExCel dressing in conjunction with a class II multilayer compression wrap and standard debridement
  Interventions: Biological: AmnioExCel dressing and compression therapy

INTERVENTIONS:
Biological: AmnioExCel dressing and compression therapy — Use of a dehydrated human amnion membrane as a biologic adjunct to the standard of care in patients with venous leg ulcers
  Arms: AmnioExCel dressing
Procedure: SOC alginate dressing and compression therapy — Alginate dressing is an absorbent wound care product that contains sodium and calcium fibers to absorb fluids and promote healing
  Arms: SOC alginate dressing

SUMMARY:
The purpose of this study is to evaluate and compare healing characteristics, reduction in the size of the wound and to measure complete healing of the wound following the application of a biologic product dressing instead of the alginate dressing along with standard debridement and compression therapy versus the standard of care treatment for VLUs. The biologic product that will be used in this study is called AmnioExCel™.

DETAILED DESCRIPTION:
Approximately 40 participants will be enrolled in this study at the Greenville Health System. Participation is anticipated to last up to 15 weeks and will include a two week screening period, randomization (Visit 1) and office visits at the study doctor's office once every week for up to 12 weeks (Visit 2 - Visit 12). All participants will receive the standard of care wound treatment during the 2 week screening period. The treatment plan outlined in treatment group 1 or treatment group 2 will be followed after randomization.

Participants will be randomly assigned (like flipping a coin) into one of two treatment groups. There is an equal chance to be enrolled into either of the two treatment groups. Neither the participant nor the study doctor can control the group assignment.

Treatment Group 1: participants will receive the standard of care treatment including the use of a multi-layer compression wrap for their VLU.

Treatment Group 2: participants will receive the application of the biologic product AmnioExCel™ dressing instead of the application of an alginate dressing in addition to standard debridement and the use of a multi-layer compression wrap for their VLU. If participants have more than one VLU, only one will be enrolled in the study and will receive the application of the AmnioExCel™ dressing. The remaining VLUs will receive the application of the alginate dressing.

AmnioExCel™ is a human cellular and tissue based product that is registered with the United States Food and Drug Administration (FDA). It is intended for use as a wound covering and is made of a dehydrated human amniotic membrane (innermost layer of the placenta) that was obtained from donated human placenta. The use of AmnioExCel™ specifically for this study is not considered as standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older
2. At least one VLU with a total surface area between 2 cm2 and 100 cm2
3. VLU present for at least 1 month
4. Presence of a VLU extending through the full thickness of the skin but not down to muscle, tendons, or bones
5. Ulcer has a clean, granulating base with minimal adherent slough
6. VLU has been treated with compression therapy for at least 14 days
7. The study VLU has < 30% area reduction with SOC treatment for the duration ≥ 2 weeks screening period
8. At least one of the following within the last 6 months:

   * An Ankle-Brachial Index (ABI) of > 0.75
   * Dorsalis Pedis (DP) systolic pressure ≥ 80 mm Hg for diabetic patients or ≥ 60 mm Hg for non-diabetic patients on study limb
   * Posterior Tibial (PT) systolic pressure ≥ 80 mm Hg for diabetic patients or ≥ 60 mm Hg for non-diabetic patients on study limb
   * Great toe systolic pressure ≥ 40 mm Hg
9. Willingness to comply with the protocol, attend all follow-up visits, complete all protocol related assessments and provide informed consent

Exclusion Criteria:

1. Presence of an active infection of the skin on the target limb such as cellulitis requiring antibiotics
2. Ulcer caused by a medical condition other than venous insufficiency
3. Ulcer suspicious for cancer
4. Known history of AIDS or HIV
5. Previously treated with tissue engineered materials (e.g., Apligraft, Dermagraft or EpiFix) or other scaffold materials (e.g., Oasis or Puraply) in the past three months on the target VLU.
6. Receipt of a biologic agent, growth factor or skin substitute within the prior 30 days
7. Known sensitivity to ethanol
8. Uncontrolled diabetes mellitus with a HgBA1c of > 10% within the past 3 months
9. Rheumatoid arthritis
10. Significant lower extremity arterial occlusive disease that would preclude the use of compression therapy
11. NYHA Class III and IV congestive heart failure (CHF)
12. Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus
13. Currently receiving radiation therapy or chemotherapy
14. Receiving immune modulators
15. Currently pregnant or trying to get pregnant
16. Breast feeding
17. Not willing to provide written informed consent or remain in compliance with the study protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Oliver, MD, Principal Investigator — Prisma Health
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from participants who sign consent will be sent in a de-identified fashion to Clemson University for data analysis. Clemson University will submit safety information to BioDLogics, LLC, in a de-identified fashion as appropriate.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC Alginate Dressing | AmnioExCel Dressing
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC Alginate Dressing | AmnioExCel Dressing | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — age, continuous
  years | 52 | 70 | 61 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Area
Description: Average percent change in wound area, computed with respect to wound area at time "0". Wound area assessed at baseline (time 0) and then weekly; change from baseline to 12 weeks reported.
Time Frame: 12 weeks
Measure: Number; unit: percentage of change
Arm/Group | SOC Alginate Dressing | AmnioExCel Dressing
Number analyzed (Participants) | 1 | 1
percentage of change | 2.94 | -31.58

2. Secondary Outcome: Change in Patient Pain Score
Description: Pain assessed at weekly visits using the Wong-Baker FACES (Family And Caregiver Education & Support) Pain Scale. Change from baseline to 12 weeks reported.
  Self-report measure of pain from 0 to 10, with higher values representing a worse outcome.
  0 = "No hurt" and 10 = "Hurts Worst"
Time Frame: 12 weeks
Measure: Number; unit: percent of change
Arm/Group | SOC Alginate Dressing | AmnioExCel Dressing
Number analyzed (Participants) | 1 | 1
percent of change | -100 | -100

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | SOC Alginate Dressing | AmnioExCel Dressing
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Alginate Dressing (N=1) | AmnioExCel Dressing (N=1)
contralateral leg venous ulcer infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Contralateral leg venous ulcer noted during office visit. Culture obtained and results were positive for infection. Pt was prescribed antibiotics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02929056/Prot_SAP_000.pdf